CLINICAL TRIAL: NCT07024121
Title: Assessing the Socio-Psychological Determinants of Sagittal Balance - PSYPOS2
Brief Title: Assessing the Socio-Psychological Determinants of Sagittal Balance
Acronym: PSYPOS 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2023/59
Record Dates: First submitted 2024-10-14; First posted 2025-06-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Healthy Spine; Posture; Sagittal Balance; Socio-Psychological Factors
Keywords: Sagittal Balance; Socio-Psychological Factors; Postural Alignment; EOS Radiography; Orthopaedic Surgery; Healthy Spine; Spinal Function; Psychological Dimensions; Spinal Radiographs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient consulting in spine surgery (Experimental): Patient consulting in spine surgery who have undergone or will undergo an EOS X-ray as part of their care pathway (particularly as part of a pre-operative assessment for hip arthroplasty) :
  Interventions: Diagnostic Test: Patient consulting in spine surgery

INTERVENTIONS:
Diagnostic Test: Patient consulting in spine surgery — Self-administered questionnaire quality of life scales

SUMMARY:
The research focuses on describing the association between socio-psychological factors, collected through standardized self-questionnaires, and the postural alignment of patients without spinal pathology consulting in the orthopaedic surgery department, as evaluated on EOS® radiographic images. This mono-centric, analytical, non-interventional, cross-sectional epidemiological study has for primary outcome to explore the relationship between socio-psychological factors and posture in patients with a healthy spine.

DETAILED DESCRIPTION:
* This study investigates the association between socio-psychological factors, collected through standardized self-questionnaires, and the postural alignment of patients without spinal pathology consulting in the orthopaedic surgery department, as evaluated on EOS® radiographic images. This mono-centric, analytical, non-interventional, cross-sectional epidemiological study has for primary outcome to explore the relationship between socio-psychological factors and posture in patients with a healthy spine.
* Posture, or sagittal balance, is a key aspect of spinal function. Considering sagittal balance is essential because its alteration leads to a decrease in quality of life and can quickly become a source of disability. Its analysis is conducted using defined parameters on spinal radiographs and is crucial for understanding spinal pathologies. Links between low back pain and posture have already been clearly reported, as well as between low back pain and socio-psychological factors. There is also evidence in the literature suggesting a relationship between socio-psychological factors and sagittal balance but these data are rare and fragmented, even though this association could be particularly pronounced in patients with spinal pathologies requiring surgical intervention.

However, it seems worthwhile to investigate this association between posture and socio-psychological characteristics in patients without spinal pathology to understand the link with other confounding or intermediate factors.

Furthermore, this association could be responsible for some of the variability in clinical and radiological outcomes of treatments, particularly surgical ones, with the presence of poor postoperative clinical outcomes despite adequate restoration of sagittal balance.

o This analytical, non-interventional study requires only one scheduled consultation within the care pathway of patients without spinal pathology consulting in the orthopaedic surgery department of the University Hospital of Bordeaux and undergoing EOS radiography as part of their care pathway. During this consultation, radiographic data and questionnaire responses will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient consulting at the investigational center (orthopaedic surgery department of Bordeaux University Hospital) who has undergone or will undergo an EOS® radiography as part of their treatment pathway (particularly in the context of a preoperative assessment for hip arthroplasty).
* Affiliation with a medical insurance scheme under the French National Health Insurance.

Exclusion Criteria:

* Spinal fusion at any operated level,
* Active or non-active spinal infection at any level,
* Spinal fracture at any level,
* Spinal deformity:

  * Scheuermann's disease (at least 3 adjacent vertebrae with wedge deformity and kyphosis increased by 5 degrees),
  * Scoliosis (Cobb angle > 10 degrees and vertebral rotation).
* History of Parkinson's disease
* Active cancer or hematologic disorder with bone involvement
* Any condition preventing the ability to respond to questionnaires with discernment
* Neurological deficit requiring urgent surgical intervention
* Hyperalgesic condition requiring urgent surgical intervention
* Polytrauma with organ failure
* Patient unable to understand study-related information
* Patient under guardianship or curatorship,
* Persons deprived of liberty by judicial or administrative decision,
* Persons receiving psychiatric care under constraint,
* Persons under guardianship,
* Patient not affiliated with a social protection scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between Global Tilt and socio-psychological variables | Baseline
  The relationship between sagittal balance, assessed using EOS® imaging and measured by the angle known as Global Tilt (GT), and socio-psychological variables .
  Sagittal balance is normal if the Global Tilt angle is less than 23.2 degrees. When the Global Tilt angle is more than 33.7 degrees, it is considered that there is a moderate pathological imbalance of the sagittal balance

SECONDARY OUTCOMES:
Correlation between sagittal balance and BBQ questionnaire | Baseline
  Correlation between other parameters of sagittal balance (T1-pelvic angle, T1 slope, LL, PT, SVA) and various psychological dimensions studied per the BBQ questionnaire BBQ : Back Belief Questionnaire : Relatively easy to implement (14 questions, ranging from 0 to 5) The Back and Belief Questionnaire (BBQ) is a standardized questionnaire with 14 items that allows for a score to be established on the extent of false beliefs held by subjects.
Correlation between sagittal balance and SF-36 | Baseline
  Correlation between other parameters of sagittal balance (T1-pelvic angle, T1 slope, LL, PT, SVA) and perceived health parameters (SF-36) SF-36v2® Health Survey : Benchmark score, validated by the scientific community.
  36 items divided into 8 dimensions. Quick (less than 10 minutes).
Relation between sagittal balance and demographic variables | Baseline
  Relation between other parameters of sagittal balance and measured demographic variables (age, sex, weight, size, diplomas, profession, ...)
Correlation between sagittal balance and TSK questionnaire | Baseline
  Correlation between other parameters of sagittal balance (T1-pelvic angle, T1 slope, LL, PT, SVA) and various psychological dimensions studied per the TSK questionnaire TSK : Tampa Scale of Kinesiophobia : Validated for low back pain and in French.
  Relatively easy to implement (17 questions, the patient must respond by choosing a number between 1 (strongly disagree) and 4 (strongly agree).
  A score above 40 indicates a patient with significant kinesiophobia..
Correlation between sagittal balance and PCS questionnaire | Baseline
  Correlation between other parameters of sagittal balance (T1-pelvic angle, T1 slope, LL, PT, SVA) and various psychological dimensions studied per the PCS questionnaire
  The Catastrophism Pain Catastrophising Scale (PCS) considers both catastrophizing thoughts and behaviors, described as a catastrophizing of pain.
  Validated in low back pain. Easy to implement (13 questions, with scores ranging from 0 to 4). Adapted into French using the PCS-CF. A score > 30 indicates a high level of catastrophizing.
Correlation between sagittal balance and HADS questionnaire | Baseline
  Correlation between other parameters of sagittal balance (T1-pelvic angle, T1 slope, LL, PT, SVA) and various psychological dimensions studied per the HADS questionnaire Hospital Anxiety and Depression Scale (HADS) questionnaire is Easy to implement (14 questions, divided between questions on anxiety and depression).
  Good internal consistency in spinal pathology Validated in French A score ≥ 11 indicates the presence of anxiety or depressive symptoms.
Correlation between sagittal balance and MSPQ questionnaire | Baseline
  Correlation between other parameters of sagittal balance (T1-pelvic angle, T1 slope, LL, PT, SVA) and various psychological dimensions studied per the MSPQ questionnaire Modified Somatic Perception Questionnaire (MSPQ) questionnaire is Easy to implement (13 questions, ranging from 0 to 3 points) Validated in spinal pathologies. The threshold has not been validated. We will use Balansyan's study as a guide, which determined that a score above 18 points appears appropriate for identifying somatic symptoms.
  This threshold has a sensitivity of 29% with very few false positives.
Correlation between sagittal balance and Big Five Inventory questionnaire | Baseline
  Correlation between other parameters of sagittal balance (T1-pelvic angle, T1 slope, LL, PT, SVA) and various psychological dimensions studied per the Big Five Inventory questionnaire Big Five Inventory - 10-questions short form is Easy to implement (10 questions).
  Short form of the Big Five Inventory validated in French. Reproducible and validated tool. Describes patients according to 5 categories: Extraversion, Agreeableness, Conscientiousness, Neuroticism, and Openness.
  The score provides percentages for each category, indicating the patient's strengths and weaknesses.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BOUYER, PROF, Principal Investigator — University Hospital, Bordeaux